CLINICAL TRIAL: NCT00092183
Title: A Randomized, Double-Blind, Parallel-Group Study Conducted Under In-House Blinding Conditions to Determine the Efficacy and Tolerability of Aprepitant for the Prevention of Chemotherapy-Induced Nausea and Vomiting Associated With Moderately Emetogenic Chemotherapy
Brief Title: An Investigational Drug for the Prevention of Chemotherapy-Induced Nausea and Vomiting (MK-0869-071)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0869-071; MK0869-071; 2004_063
Record Dates: First submitted 2004-09-21; First posted 2004-09-24 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Nausea; Vomiting; Breast Neoplasms
Keywords: Chemotherapy-Induced Nausea and Vomiting
MeSH Terms: conditions — Nausea; Vomiting; Breast Neoplasms | interventions — Aprepitant; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0869, aprepitant / Duration of Treatment: 3 days
Drug: Comparator: ondansetron / Duration of Treatment: 3 days

SUMMARY:
This protocol will study an investigational drug treatment plan against standard therapy in the prevention of chemotherapy-induced nausea and vomiting in patients diagnosed with breast cancer who are to be treated with up to 4 cycles of non-cisplatin moderately emetogenic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of breast cancer requiring treatment with non-cisplatin moderately emetogenic chemotherapy.

Exclusion Criteria:

* Patient has a central nervous system malignancy.
* Patient will receive radiation to the abdomen or pelvis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 866 (Actual)
Dates: Start 2002-10-10 (Actual); Primary Completion 2003-12-01 (Actual); Study Completion 2004-02-11 (Actual)

PRIMARY OUTCOMES:
Emesis and use of rescue medication
Safety and tolerability

SECONDARY OUTCOMES:
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Warr DG, Hesketh PJ, Gralla RJ, Muss HB, Herrstedt J, Eisenberg PD, Raftopoulos H, Grunberg SM, Gabriel M, Rodgers A, Bohidar N, Klinger G, Hustad CM, Horgan KJ, Skobieranda F. Efficacy and tolerability of aprepitant for the prevention of chemotherapy-induced nausea and vomiting in patients with breast cancer after moderately emetogenic chemotherapy. J Clin Oncol. 2005 Apr 20;23(12):2822-30. doi: 10.1200/JCO.2005.09.050. PMID 15837996
- Available data/document: CSR Snyopsis — http://www.merck.com/clinical-trials/policies-perspectives.html